CLINICAL TRIAL: NCT03765957
Title: Clinical Research on Treatment of Psoriasis by Human Umbilical Cord-derived Mesenchymal Stem Cells
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Yijing He, Associate professor, Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-MSC/CSU/PS
Record Dates: First submitted 2018-08-28; First posted 2018-12-05 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Psoriasis
Keywords: Mesenchymal Stem Cells
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesenchymal Stem Cells (Experimental): The mesenchymal stem cells will be derived from human umbilical cord. After the subjects are screened and qualified, random number envelopes will be selected to group 12 subjects into group A, group B, group C and group D at a ratio of 1:1:1:1. The subjects of group A and B will be injected intravenously with 1.5x10E6/kg and 2.0x10E6/kg（according to the weight of subject）mesenchymal stem cells respectively at baseline and every 2 weeks, 4 times is a course of treatment. Subjects will be followed up for evaluation on 15 days, 30 days, 45 days, month 2, month 3 and month 6 after treatment. The subjetcts of group C and D will be injected intravenously with 2.5x10E6/kg and 3.0x10E6/kg （according to the weight of subject）mesenchymal stem cells respectively at baseline and every 4 weeks, 2 times is a course of treatment. Subjects will be followed up for evaluation on 15 days, 30 days, 45 days, month 2, month 3 and month 6 after treatment.
  Interventions: Biological: Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — After the subjects are screened and qualified, random number envelopes will be selected to group 12 subjects into group A, group B, group C and group D at a ratio of 1:1:1:1. The subjetcts of group A and B will be injected intravenously with 1.5x10E6/kg and 2.0x10E6/kg（according to the weight of subject）mesenchymal stem cells respectively at baseline and every 2 weeks, 4 times is a course of treatment. Subjects will be followed up for evaluation on 15 days, 30 days, 45 days, month 2, month 3 and month 6 after treatment. The subjetcts of group C and D will be injected intravenously with 2.5x10E6/kg and 3.0x10E6/kg （according to the weight of subject）mesenchymal stem cells respectively at baseline and every 4 weeks, 2 times is a course of treatment. Subjects will be followed up for evaluation on 15 days, 30 days, 45 days, month 2, month 3 and month 6 after treatment. Besides MSCs, moisturizers such as boric acid ointment will be given to all subjects.
  Other Names: Human Umbilical Cord-derived Mesenchymal Stem Cells

SUMMARY:
To evaluate the effect and safety of treatment of psoriasis by human umbilical cord-derived mesenchymal stem cel

DETAILED DESCRIPTION:
Psoriasis is a chronic and recurrent inflammatory skin disease and its histological features are characterized by epidermal hyperplasia, increased angiogenesis and immune cell infiltration. Psoriasis prevalence is about 0.1%-3%, affecting approximately 125 million people worldwide. In China, there are about 10 million psoriasis patients.

Human umbilical cord-derived MSC (huc-MSC) has many advantages for the treatment of immune disease. Because it was demonstrated that huc-MSCs are effective in modulating immune cells and treating diseases and it has low immunogenicity. Furthermore, huc-MSCs do not raise ethical issue for clinical applications.

Some experimental results and cases has showed that mesenchymal stem cell (MSC) can prevent or treat psoriasis. This clinical study is conducted to provide more data to evaluate the effect and safety of treatment of psoriasis by human umbilical cord-derived mesenchymal stem cell.

ELIGIBILITY:
Inclusion Criteria:

1.Understanding the whole process of the study, voluntary participation and signed the informed consent; 2.18 Years to 65 Years old, Body Mass Index (BMI) between 18.5-35; 3.Diagnosed according to biopsy for Psoriasis vulgaris for more than 6 months and resistance to phototherapy, systemic therapy, or a combination of these therapies,BSA(body surface area)>10%, PGA≥3 and PASI>10 at baseline; 4. Patients participated in any stem cell therapy within 6 months;

Exclusion Criteria:

1. WBC(white blood cell count ) <3.5x109/L, blood platelet count<100x109/L, hemoglobin<100g/L serum creatinine>1.5 x ULN(upper limit of normal), bilirubin > 1.5 x ULN(upper limit of normal), AST(SGOT,glutamic-oxalacetic transaminase)/ALT(SGPT,glutamic-pyruvic transaminase) >2.0 x ULN(upper limit of normal);Either HIV-antibody(human immunodeficiency virus-antibody), HBV-antibody (hepatitis B virus-antibody ) or syphilis antibody is positive;
2. Have a serious heart, lung, kidney and other vital organs and endocrine system lesions and the history,Patients suffering from any acute or chronic infectious diseases, patients suffering from malignant tumor; Mental disorders, history of alcohol abuse, drug or other substance abuse;
3. Patients who have received systemic therapy within recent one month or topical therapy in two weeks;
4. Having a serious allergic history or being allergic to two or more than 2 kinds of food or drugs;
5. Pregnant women, or women who ready for pregnancy or lactating; Patients participated in any clinical trials within 3 months; Other cases which researchers believe that can not enroll.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Achieving Psoriasis Area and Severity Index ≥75% (PASI 75) Improvement | Month 6
  The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation (scaling), erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease. Participants achieving PASI 75 was defined as having an improvement of at least 75% in the PASI scores compared to baseline.
Number of Participants Achieving a Physician Global Assessment (PGA) of (0, 1) | Month 6
  The PGA is a physician's determination of the participant's psoriasis lesions overall categorized by descriptions for induration, erythema, and scaling.

SECONDARY OUTCOMES:
Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score | Baseline, Month 6
  The DLQI is a simple, participant-administered, 10 question, validated, quality-of-life questionnaire that covers 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." Totals range from 0 to 30 (less to more impairment), and a 5 point change from baseline is considered clinically relevant. Least Square (LS) Means in total DLQI score were calculated using Mixed Model Repeated Measures (MMRM) with baseline score as covariate, treatment, pooled center, visit and treatment-by-visit interaction as fixed effects.
Adverse event | Baseline, Month 6
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Chen, M.D. Ph.D, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Comella K, Parlo M, Daly R, Dominessy K. First-in-man intravenous implantation of stromal vascular fraction in psoriasis: a case study. Int Med Case Rep J. 2018 Mar 21;11:59-64. doi: 10.2147/IMCRJ.S163612. eCollection 2018. PMID 29606893
- [Background] Lee YS, Sah SK, Lee JH, Seo KW, Kang KS, Kim TY. Human umbilical cord blood-derived mesenchymal stem cells ameliorate psoriasis-like skin inflammation in mice. Biochem Biophys Rep. 2016 Oct 8;9:281-288. doi: 10.1016/j.bbrep.2016.10.002. eCollection 2017 Mar. PMID 28956015
- [Background] Boehncke WH, Schon MP. Psoriasis. Lancet. 2015 Sep 5;386(9997):983-94. doi: 10.1016/S0140-6736(14)61909-7. Epub 2015 May 27. PMID 26025581
- [Background] Owczarczyk-Saczonek A, Krajewska-Wlodarczyk M, Kruszewska A, Placek W, Maksymowicz W, Wojtkiewicz J. Stem Cells as Potential Candidates for Psoriasis Cell-Replacement Therapy. Int J Mol Sci. 2017 Oct 20;18(10):2182. doi: 10.3390/ijms18102182. PMID 29053579
- [Background] Guan LX, Guan H, Li HB, Ren CA, Liu L, Chu JJ, Dai LJ. Therapeutic efficacy of umbilical cord-derived mesenchymal stem cells in patients with type 2 diabetes. Exp Ther Med. 2015 May;9(5):1623-1630. doi: 10.3892/etm.2015.2339. Epub 2015 Mar 9. PMID 26136869
- [Background] Ra JC, Kang SK, Shin IS, Park HG, Joo SA, Kim JG, Kang BC, Lee YS, Nakama K, Piao M, Sohl B, Kurtz A. Stem cell treatment for patients with autoimmune disease by systemic infusion of culture-expanded autologous adipose tissue derived mesenchymal stem cells. J Transl Med. 2011 Oct 21;9:181. doi: 10.1186/1479-5876-9-181. PMID 22017805
- [Background] Dahbour S, Jamali F, Alhattab D, Al-Radaideh A, Ababneh O, Al-Ryalat N, Al-Bdour M, Hourani B, Msallam M, Rasheed M, Huneiti A, Bahou Y, Tarawneh E, Awidi A. Mesenchymal stem cells and conditioned media in the treatment of multiple sclerosis patients: Clinical, ophthalmological and radiological assessments of safety and efficacy. CNS Neurosci Ther. 2017 Nov;23(11):866-874. doi: 10.1111/cns.12759. Epub 2017 Sep 29. PMID 28961381
- [Background] Cui GH, Wang YY, Li CJ, Shi CH, Wang WS. Efficacy of mesenchymal stem cells in treating patients with osteoarthritis of the knee: A meta-analysis. Exp Ther Med. 2016 Nov;12(5):3390-3400. doi: 10.3892/etm.2016.3791. Epub 2016 Oct 11. PMID 27882169
- [Derived] Cheng L, Wang S, Peng C, Zou X, Yang C, Mei H, Li C, Su X, Xiao N, Ouyang Q, Zhang M, Wang Q, Luo Y, Shen M, Qin Q, Wang H, Zhu W, Lu G, Lin G, Kuang Y, Chen X. Human umbilical cord mesenchymal stem cells for psoriasis: a phase 1/2a, single-arm study. Signal Transduct Target Ther. 2022 Aug 5;7(1):263. doi: 10.1038/s41392-022-01059-y. PMID 35927231